CLINICAL TRIAL: NCT00823849
Title: A Randomized, Control,Open Label, Multicentre Clinical Study to Evaluate the Efficacy and Safety of Cilostazol and Probucol Alone and in Combination on Atherosclerosis Related Biomarker
Brief Title: Study of Cilostazol and Probucol to Assess Their Effects on Atherosclerosis Related Biomarker
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Otsuka Beijing Research Institute (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 246-08-802-01
Record Dates: First submitted 2009-01-14; First posted 2009-01-16 (Estimated); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Type 2 Diabetes Mellitus; Arteriosclerosis Obliterans
Keywords: type 2 diabetes mellitus, with Arteriosclerosis obliterans
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Arteriosclerosis Obliterans | interventions — Cilostazol; Probucol; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental)
  Interventions: Drug: Cilostazol
- 2 (Experimental)
  Interventions: Drug: Probucol
- 3 (Experimental)
  Interventions: Drug: Cilostazol+Probucol
- 4 (Other): Control Group, regular treatment
  Interventions: Other: Control Group

INTERVENTIONS:
Drug: Cilostazol — From 50mg, Bid, PO after breakfast and dinner. After 1-week of administration, if no significant study drug related discomfort, the dose can increase to 100mg, Bid, PO. Otherwise, remain at the 50 mg level.
  Other Names: pletaal
  Arms: 1
Drug: Probucol — 250 mg Bid, PO after breakfast and dinner.
  Other Names: Changtai
  Arms: 2
Drug: Cilostazol+Probucol
  Other Names: Pletaal and Changtai
  Arms: 3
Other: Control Group — Routine treatment
  Other Names: Routine treatment
  Arms: 4

SUMMARY:
1. To evaluate the efficacy of Cilostazol and Probucol alone and in combination on atherosclerosis related biomarker
2. To evaluate the safety of Cilostazol and Probucol alone and in combination on atherosclerosis related biomarker

DETAILED DESCRIPTION:
Efficacy evaluation:

Primary efficacy index:

After 12 weeks of treatment, the change of arteriosclerosis related biomarker in 4 modality groups, comparing with the base line information

Secondary efficacy index:

After 8 weeks of treatment, the change of arteriosclerosis related biomarker in 4 modality groups, comparing with the base line information

Safety evaluation:

1. Adverse Event
2. Vital Sign and Physical Examination
3. 12-lead ECG
4. Laboratory Tests (including blood routine examination, routine urine analysis, blood biochemistry examination, glycosylated hemoglobin)

ELIGIBILITY:
Inclusion Criteria:

* 40~75-year-old male or female
* Clarified diagnosis of type 2 diabetes mellitus
* Arteriosclerosis obliterans (ASO) is diagnosed (ASO diagnoses should meet at least one of the conditions as below:

  * ABI<1.0;
  * The pulse of popliteal artery or dorsalis pedis artery is weeken significantly or is different between left and right sides
  * Intermittent claudication, diagnosed as ASO by doctor
  * Ultrasonogram showed that there was atherosclerotic plaque in lower limb within 1 year
* Informed Consent Form Signature

Exclusion Criteria:

* Has an allergic history to study drugs
* Use one of the following drugs: other antiplatelet or anticoagulation agents except Aspirin, other hypolipidemic agents except Statins
* Type 1 diabetes mellitus, specific diabetes mellitus, or gestational diabetes mellitus
* Has severe ASO above Fontaine IIb,
* Hemorrhagic tendency or hemorrhagic disease (such as gastrointestinal tract hemorrhage, etc.)
* Had a myocardial infarction, angina pectoris, or cerebral infarction within the last 3 months
* Congestive heart failure
* Is pregnant, or potentially pregnant, or breastfeeding
* Severe hepatic insufficient or severe renal insufficiency (AST or ALT is 2.5 times higher than the upper limit of the normal value range, or serum creatinine is 1.2 times higher than the upper limit of the normal value range)
* Persistent or hardly controlled hypertension (such as malignant hypertension, BP> 160/100 mmHg)
* Severe ventricular arrhythmia (such as multiple and multifocal premature ventricular contractions)
* Has a medical history that includes a cardiac syncope or a primary syncope
* Has conditions that may prolong QT interval (such as congenital long QT syndrome, taking drugs which prolong QT interval, hypokalemia or hypomagnesemia, etc.)
* Has severe complications (such as diabetes mellitus ketoacidosis, nonketotic hyperosmolar diabetic coma, malignant tumor, severe anaemia, severe hematologic diseases, etc.)
* Other conditions that would exclude the subject from this study by doctor's judgement

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2008-10; Primary Completion 2009-08 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Primary Efficacy Evaluation: Comparing with the basic line information, the change value of arteriosclerosis related biomarker in 4 groups after 12 weeks of treatment. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohui Guo, M.D., Principal Investigator — No 1 Hospital of Peking University
Locations (1):
- Peking University First Hospital, Beijing, China